CLINICAL TRIAL: NCT00968760
Title: CD19-specific T Cell Infusion in Patients With B-Lineage Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Alaunos Therapeutics (Industry); Intrexon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0635; 5R01CA141303-03 (NIH); NCI-2011-01129 (Registry Identifier: NCI CTRP); RP120241 (Other Grant/Funding Number: CPRIT)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma; B-cell Lymphoma
Keywords: CD19+ lymphoid malignancies; non-Hodgkin's Lymphoma; NHL; small lymphocytic lymphoma; SLL; follicular lymphoma; mantle cell lymphoma; gene cell transfer; CD19-specific T cells; Stem Cell Transplant; T Cell Infusion; Chemotherapy; Leukapheresis; BCNU; carmustine; Cytarabine; Etoposide; Interleukin-2; Proleukin; Melphalan; Rituximab; T cell therapy
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Leukapheresis; Stem Cell Transplantation; Interleukin-2; aldesleukin; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CD19-specific T cell Infusion without IL-2 (Experimental): Conditioning Regimen of Chemotherapy (Carmustine, Cytarabine, Etoposide, and Melphalan), Stem Cell Transplant, and Gene Transfer
  Group 1 - low dose of T cells without IL-2.
  Group 3 - higher dose of T cells without IL-2.
  Interventions: Procedure: Leukapheresis; Procedure: Stem Cell Transplant; Procedure: CD19-specific T Cell Infusion; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan
- CD19-specific T cell Infusion with IL-2 (Experimental): Conditioning Regimen of Chemotherapy (Carmustine, Cytarabine, Etoposide, and Melphalan), Stem Cell Transplant, and Gene Transfer
  Group 2 - higher dose of T cells with IL-2.
  Group 4 - higher dose of T cells with IL-2.
  Interventions: Procedure: Leukapheresis; Procedure: Stem Cell Transplant; Procedure: CD19-specific T Cell Infusion; Drug: IL-2; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan

INTERVENTIONS:
Procedure: Leukapheresis — Leukapheresis #1 - For Collecting T Cells
  Leukapheresis #2 - For Collecting Stem Cells, month following #1
  Blood drawn through vein, passed through a machine to collect specific blood cells, then remaining blood returned, about 3 hours to complete.
Procedure: Stem Cell Transplant — Stem cell infusion by vein over 30-45 minutes on Day 0
  Other Names: SCT
Procedure: CD19-specific T Cell Infusion — T Cell Infusion (Gene Transfer) by vein over 15-30 minutes sometime between Day +2 through Day +7.
Drug: IL-2 — Group 2 or 4, IL-2 dose of 0.3 x 10^6 U/m^2 injected under skin, once a day for up to 14 days; first dose on day of T cell infusion.
  Other Names: Interleukin-2; Proleukin
  Arms: CD19-specific T cell Infusion with IL-2
Drug: Carmustine — 300 mg/m^2 IV over 1 hour on Day -6
  Other Names: BCNU; BiCNU
Drug: Etoposide — 200 mg/m^2 IV over 3 hours every 12 hours on Days -5 to -2
  Other Names: VePesid
Drug: Cytarabine — 200 mg/m^2 by vein over 1 hour every 12 hours on Days -5 to -2.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Melphalan — 140 mg/m^2 IV over 30 minutes on Day -1
  Other Names: Alkeran

SUMMARY:
Sometimes researchers change the DNA (genetic material in cells) of donated T cells (white blood cells that support the immune system) using a process called "gene transfer." Gene transfer involves drawing blood from the patient, and then separating out the T-cells using a machine. Researchers then perform a gene transfer to change the T-cells' DNA, and then inject the changed T-cells into the body of the patient.

The goal of this clinical research study is to learn if an investigational type of gene transfer can be given reliably and safely in patients with advanced B-cell lymphoma. B cells are a type of white blood cell that fights infection and disease. Lymphoma is a type of cancer that affects the immune system, including B cells.

The gene transfer involves drawing blood, separating out T cells (white blood cells that fight infection and disease), changing the T cells' DNA (genetic material) in a specific way, and returning the changed T cells back to the body.

Researchers want to learn the highest dose of the changed T cells that can be given safely. Researchers also want to learn how long the changed T cells remain in the participant's body, and if the changed T cells can reliably treat B-cell lymphoma. Finally, researchers want to learn if interleukin-2 (IL-2) can help the changed T cells last longer in the body.

DETAILED DESCRIPTION:
Study Plan:

This study has 3 steps: chemotherapy, a stem cell transplant, and gene transfer. If the disease relapses (returns) during the study, you may receive the T-cell infusion without having a stem cell transplant. Your study doctor will decide if you will receive the stem cell transplant or not.

The chemotherapy combination in this study (carmustine [BiCNU®], cytarabine [Cytosar-U®], etoposide [Vepesid®], and melphalan [Alkeran®] is given to try to destroy any remaining tumor cells and prepare the body for the stem cell transplant and/or T-cell infusion.

If you receive the T cells without transplant, you may receive additional chemotherapy before the T cell infusion, if your doctor thinks it is needed. Your treating doctor will discuss these chemotherapy drugs with you, and you may sign an additional consent for those chemotherapy drugs as standard of care.

A stem cell transplant is designed to help the body attack the cancer cells that may remain after chemotherapy.

The gene transfer involves drawing blood, separating out T cells, changing the cells' DNA in the laboratory, and returning the genetically changed cells back to the body. T cells are a type of white blood cell that fight infection. The type of gene transfer being used in this study is designed to help your T cells better fight B-cell lymphoma. These genetically changed T cells are designed to fight B-cell lymphoma by targeting CD19 (a chemical "marker" that is found on certain B-cell lymphoma cells).

IL-2 (Proleukin®) is designed to help T cells grow. In this study, researchers want to learn if it can help the genetically changed T cells grow and last longer in the body.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of T cells, with or without IL-2, based on when you joined this study.

The first group of participants will receive the lowest dose of T cells. Each new group will receive a higher dose of T cells than the group before it, if no intolerable side effects were seen. Up to 4 dose combinations of T cells will be tested.

Tests Before Leukapheresis:

Before each of the 2 leukapheresis procedures (described below), the following tests and procedures will be performed:

* Blood (about 4 tablespoons) will be drawn and used for routine tests and to look for diseases such as hepatitis and HIV.
* To check your lung function, you will have breathing tests. A chest X-ray will be performed to check for infection.

Leukapheresis #1 or Standard Blood Draw (For Collecting T Cells) You will visit the Apheresis Clinic at MD Anderson to have leukapheresis performed. Leukapheresis is a procedure for removing blood from the body in order to collect specific blood cells. The remaining blood is then returned to the body.

Blood will be drawn through a needle in a vein in one arm, then passed through a machine, and then the remaining blood will be returned back to you through a needle in a vein in your other arm. The machine will remove a sample of your white blood cells. This process will take about 3 hours to complete.

Blood may also be collected through a standard blood draw. Blood (less than 7 tablespoons) containing circulating T cells will be drawn over 1-2 days using one or more needle sticks in your arm.

Your white blood cell sample will be sent to a lab at MD Anderson so the genetically modified T cell product can be made. The modified T cells will be grown in the lab.

It will take about 7 weeks to modify and grow the necessary number of genetically modified T cells. If researchers are unable to create a high enough dose of T cells for you in the lab, you will be taken off study.

Placement of Central Venous Catheter:

Before the second leukapheresis, you will receive a central venous catheter. This is a sterile flexible tube that will be placed into a large vein in your upper chest, while you are under local anesthesia. The study investigator will explain this procedure to you in more detail, and you will be required to sign a separate consent form for it.

When possible, all drugs that need to be given by vein will be given using the catheter. You will also receive the T cell product through the catheter.

Leukapheresis #2 (For Collecting Stem Cells) only in patients receiving a stem cell transplant:

About a month after your first leukapheresis, you will return to have the procedure repeated a second time. This time, the blood cells collected will be a sample of blood-forming stem cells. The stem cells will be given back to you after your chemotherapy. If a high enough number of stem cells cannot be collected, however, you will be taken off study.

A stem cell transplant is part of this study's treatment plan, but in some cases, participants in this study will have their stem cells collected as part of another research study or for routine care.

Chemotherapy and Stem Cell Transplant:

After your stem cells have been successfully collected, you will be admitted to the hospital to receive chemotherapy. You will stay in the hospital for about 3-4 weeks.

* On Day 1, you will receive carmustine by vein over 1 hour.
* Every 12 hours on Days 2-5, you will receive cytarabine by vein over 1 hour and etoposide by vein over 3 hours.
* On Day 6, you will receive melphalan by vein over 30 minutes.
* On Day 7, the stem cells that were collected earlier will be given back to you ("transplanted") by vein over 30-45 minutes. Day 7 is also called Day 0, since it is the day of the transplant. The days after the transplant are called Days +1, +2, and so on.

After the stem cell transplant, the study investigator will decide if you are still eligible to receive the T cell infusion (and IL-2, if you are assigned to receive it). If you have any infections or intolerable side effects, or if you are taking certain types of steroids by mouth or injection, you will be taken off study. If you do not receive the T cell infusions, you would not need to return for the follow-up described below.

If you have had prior involvement of disease in your brain/spine area, your physician may give you a different chemotherapy regimen consisting of the following:

* On Day 1, you will receive carmustine by vein over 1 hour.
* Every 12 hours on Days 2-3, you will receive thiotepa by vein over 1 hour
* On Day 7, the stem cells that were collected earlier will be given back to you ("transplanted") by vein over 30-45 minutes. Day 7 is also called Day 0, since it is the day of the transplant. The days after the transplant are called Days +1, +2, and so on.

T Cell Infusion (Gene Transfer):

You will receive the T cell infusion sometime between Day +2 through Day +7. (The exact day will be as soon as you are eligible.) The T cell infusion will be given by vein over 15-30 minutes. The infusion may be divided into two parts at least 24 hours apart. The first part of the infusion will be a much smaller part to ensure that you have no immediate side effects. During the infusion, your vital signs will be checked.

Alternatively, your doctor may decide that it is better for you to receive the infusion on one day by vein over 15-30 minutes. During the infusion, your vital signs will be checked.

Before the T cell infusion, you will receive drugs to lower your risk of allergic reaction to the T cells. Acetaminophen (Tylenol®) will be given by mouth, and diphenhydramine (Benadryl®) will be given by vein over a few minutes.

IL-2 Administration:

If you are in Group 2 or 4, IL-2 will be injected under the skin, once a day for up to 14 days. The first dose will be on the day of your T cell infusion.

Before each IL-2 injection, you will receive drugs to lower your risk of allergic reaction to the IL-2. Acetaminophen will be given by mouth. Diphenhydramine will be given by mouth or by vein over a few minutes.

Study Tests:

Every day while you are in the hospital, blood (about 2 teaspoons) will be drawn for routine tests.

On the day of the T-cell infusion, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of vital signs and weight.
* You will be asked about any side effects you may have had.
* Your medical history will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Within 3 days, 1 week, and 2 weeks after the T cell infusion, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of vital signs and weight.
* Your medical history will be recorded.

At 1, 2, 3, 6, and 12 months (+/-5 days), blood (about 2 teaspoons each time) will be drawn for research to look for the modified T cells and to measure the number of B cells and other (non-modified) T cells. Like T cells, B cells are part of your immune system.

Follow-Up:

At about 1, 2, 3, 6, and 12 months after the stem cell transplant, you will return for follow-up visits. At each visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of vital signs and weight.
* Your medical history will be recorded.
* Blood (about 1-2 tablespoons) will be drawn for routine tests and for research to look for the modified T cells and to measure the number of B cells and other T cells. Part of the blood sample at 12 months will be tested for HAMA.
* Other tests to check your health may also be performed if needed, such as CT scans, PET/CT scans, and/or bone marrow aspirations and biopsies.

If the disease comes back or a side effect occurs during the 12 months after the stem cell transplant, you may be asked to return for additional follow-up visits as needed.

Length of Study Participation:

If you have any infections or intolerable side effects, you will be taken off study early.

If you complete the study as planned, you will be off-study after your last follow-up visit.

Request for Autopsy:

In the event of death due to any cause, an autopsy will be requested from your family if it is possible.

Long-Term Follow-Up:

For safety reasons, the U.S. Food and Drug Administration (FDA) requires patients receiving gene transfer to have long-term follow-up for at least 15 years after receiving the gene transfer. You will be asked to sign a separate consent form for long-term follow up. That study is known as Protocol 2006-0676, and the follow-up will begin 1 year after the gene transfer study.

This is an investigational study. The chemotherapy and stem cell transplant in this study are commercially available and FDA approved. The gene transfer is not commercially available or FDA approved. At this time, gene transfer is only being used in research.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of CD19+ lymphoid malignancies that are beyond first remission or primary refractory to treatment.
2. Age 18 to 75 years.
3. Zubrod performance 0-1 or Karnofsky greater than or equal to 80%.
4. Patient able to provide written informed consent.
5. Patient able to provide written informed consent for the long-term follow-up gene therapy study.
6. Eligibility at time of transplant conditioning regimen (criteria 6-13): Zubrod performance 0-1 or Karnofsky greater than or equal to 80%.
7. Left ventricular ejection fraction >/= 40%. No uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease.
8. No symptomatic pulmonary disease. FEV1, FVC and DLCO >/= 50% of expected, corrected for hemoglobin.
9. Serum creatinine </= 1.8mg/dL or creatinine clearance >/= 40 cc/min.
10. Adequate hepatic function, as defined by SGPT <3 X upper limit of normal; serum bilirubin and alkaline phosphatase <2 X upper limit of normal, or considered not clinically significant.
11. If positive Hepatitis B and/or Hepatitis C serology, discuss with Principal Investigator or designee and consider liver biopsy.
12. No pleural/pericardial effusion or ascites estimated to be >1L.
13. Not breast feeding or pregnant. Pregnancy determined by a positive beta HCG test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization.
14. Eligibility at time of T-cell infusion (criteria 14-15): No systemic corticosteroids within 3 days prior to T-cell infusion.
15. Not experiencing any new Grade >2 (CTC version 4) adverse neurologic, pulmonary, cardiac, gastrointestinal, renal or hepatic (excluding albumin) event within 24 hours prior to T-cell infusion.
16. Eligibility criteria for administration of IL-2 after T-cell infusion: Absence of new adverse event of grade >2 (CTC vs. 4) involving cardiopulmonary, hepatic (excluding albumin), gastrointestinal, neurologic, or renal toxicity probably or definitely attributed to infused T cells within one week of cells.

Exclusion Criteria:

1. Positive beta HCG in female of child-bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
2. Patients with known allergy to bovine or murine products.
3. Positive serology for HIV.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of T-cells ± IL-2 | Continuously monitored up to infusions (+14 days) then at 1 day, 3 days, 1 week, and 2 weeks after T cell infusion
  The MTD is the highest dose at which at least 6 participants treated with the proportion of participants having dose limiting toxicities (DLT) < 1/3.
  DLT is defined as a new adverse event of grade >3 involving cardiopulmonary, gastrointestinal, hepatic (excluding albumin), neurological, or renal Common Terminology Criteria for Adverse Events (CTCAE) version 4 parameters that is probably or definitely related to the infused T-cell product.

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kebriaei P, Singh H, Huls MH, Figliola MJ, Bassett R, Olivares S, Jena B, Dawson MJ, Kumaresan PR, Su S, Maiti S, Dai J, Moriarity B, Forget MA, Senyukov V, Orozco A, Liu T, McCarty J, Jackson RN, Moyes JS, Rondon G, Qazilbash M, Ciurea S, Alousi A, Nieto Y, Rezvani K, Marin D, Popat U, Hosing C, Shpall EJ, Kantarjian H, Keating M, Wierda W, Do KA, Largaespada DA, Lee DA, Hackett PB, Champlin RE, Cooper LJ. Phase I trials using Sleeping Beauty to generate CD19-specific CAR T cells. J Clin Invest. 2016 Sep 1;126(9):3363-76. doi: 10.1172/JCI86721. Epub 2016 Aug 2. PMID 27482888
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org